CLINICAL TRIAL: NCT03573921
Title: The Therapeutic Role of Gastrografin for Treating Small Bowel Obstruction in Children: A Multi-Centre Canadian Prospective Study
Brief Title: Gastrografin for Treating Small Bowel Obstruction in Children
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Poor recruitment to date.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LHSC032018
Record Dates: First submitted 2018-06-11; First posted 2018-06-29 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Small Bowel Obstruction
Keywords: Paediatrics; Gastrografin
MeSH Terms: interventions — Diatrizoate Meglumine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Clustered study, where each centre will select which of the two study arms (Gastrografin or Saline solution) they will offer at their centre.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastrografin Arm (Experimental): Patients will receive a single dose of undiluted Gastrografin via the nasogastric tube at 24 hours after admission for small bowel obstruction. The dose of Gastrografin will be proportional to the patient's weight and age and will be based off of the recommendations from the drug manufacturer. Dosages will range from 30 ml for infants to children less than 5 years old and 60 ml for children 5-18 years and will not be diluted.
  Interventions: Drug: Gastrograﬁn
- Control Arm (Experimental): Patients will receive a single dose of saline solution via the nasogastric tube at 24 hours after admission for small bowel obstruction. The volume of saline solution will be proportional to the volume of Gastrografin patients of similar weight and age would receive.
  Interventions: Other: Saline solution (control treatment)

INTERVENTIONS:
Drug: Gastrograﬁn — Patients will receive a single dose of Gastrografin via the nasogastric tube at 24 hours after hospital admission. After receiving Gastrografin, patients will receive the same standard non-surgical management that patients outside of the trial receive.
  Other Names: diatrizoate meglumine and diatrizoate sodium solution
  Arms: Gastrografin Arm
Other: Saline solution (control treatment) — Patients will receive a single dose of saline solution via the nasogastric tube at 24 hours after hospital admission. After receiving saline solution, patients will receive the same standard non-surgical management that patients outside of the trial receive.
  Arms: Control Arm

SUMMARY:
This is a multi-centre clustered open label clinical trial testing the effectiveness of adding Gastrografin to standard non-surgical management of small bowel obstruction. Gastrografin is a radiopaque contract agent that exhibits a mild laxative effective due to its high osmolarity and ability to pull water into the intestines and bowels as a lubricant. Small bowel obstruction is a mechanical or function obstruction that prevents normal bowel function. The standard treatment for small bowel obstruction is non-surgical and includes decompressing the abdomen, fluid resuscitation, nothing by mouth, and time. In some cases if non-surgical management is not effective in resolving the obstruction, surgical intervention is required. Gastrografin in addition to standard non-surgical management has been shown to reduce the rate of surgery, length of hospital stay, and time to resolution in similar clinical scenarios, such as meconium ileus and meconium plug syndrome. However, it has never been tested in children with small bowel obstruction. This study is a clustered open label study, meaning that each participating centre will select the type of treatment they will offer at their centre. The treatment options are either the Gastrografin arm (a single dose of Gastrografin plus non-surgical management) or the Control arm (a single dose of saline solution plus non-surgical management). After each group receives saline or Gastrografin they will continue with the same non-surgical treatment that patients not participating in the trial would receive. Participating in the study does not preclude the need for urgent or emergent surgical intervention and at any point in the study, if the patient requires surgery for their small bowel obstruction they will undergo surgical intervention. The outcomes of this study are the rate of surgical intervention, length of stay, time to first and full feeds, and rate of complications.

DETAILED DESCRIPTION:
This will be a 2-year multi-centre clustered open-label clinical trial examining the therapeutic use of a drug called Gastrografin in reducing the length of hospital stay, time to feeding, and rate of surgery in children with a small bowel obstruction. Each participating centre will select which of the two treatment options they will offer to patients at their centre. The patients at each centre will be aware of the treatment offered at thier centre before making the decision whether to participate in the study. The two arms of the study are: Gastrografin or Control (saline solution). If a patient declines participation in the arm offered at their centre they will not be enrolled in the study. The investigators have chosen an open-label cluster study design instead of a randomized controlled trial (RCT) because it is common for RCTs to be stopped early due to poor recruitment rates within paediatric surgery. A 2018 systematic review reported that of the 137 eligible RCTs within paediatric general surgery only 19% successfully achieved the projected recruitment number and further, only 53% of studies that provided an expected completion date achieved the target. Based on the power calculation for this study, the investigators require a total of 146 patients (73 in each group) to achieve 80% power. Therefore if a RCT design is used, estimating a typically recruitment rate of 40-50%, it would take over 8 years to reach the required sample size between the participating centres. With a prospective, open-label design, the investigators anticipate the total number of possible patients that can be approached to participate in the study across all centres to be between 152-160 patients over the two years. The investigators estimate large centres will on average recruit between 10-12 patients per year, medium centres 6-8 patients per year, and small centres 2-4 patients per year.

Consent/Assent will be obtained from the parents/caregivers prior to participation in the study. Assent, in addition to parental/caregiver consent, will be used for patients between the ages of 7 and 11. Prior to the patient participating in any study-related activities, consent will be obtained. Patients will be included in this study if they are between the ages of 6 months and 18 years of age, are diagnosed with a small bowel obstruction, and have undergone 24 hours of monitoring and non-surgical management. Patients will be excluded from the study if they have thyroid stimulating hormone or thyroxine levels outside of the normal range, are taking any thyroid replacement medication, have previously had thyroid surgery, have an allergy to the medical or non-medical ingredients in Gastrografin, and weigh less than 10kg at the time of diagnosis.

Recruitment will begin following a positive diagnosis of a small bowel obstruction secondary to previous surgery, assessment by the surgical team, and after the patient has been admitted to the hospital for a twenty-four hour period of non-surgical management, which includes nasogastric (NG) decompression, fluid resuscitation, and maintenance. The patients will be assessed by the surgical team on a regular basis during this time as part of standard care and enrollment in the study does not preclude urgent or emergent surgical intervention. After 24 hours of admission, the patient will be approached to participate in the study. The study will be explained to the patient and their parents/caregivers by the research team. The patient and their family will be given as much time as required to talk among themselves about the study and ask any questions about the study to the research team. Depending on which study arm is offered at their hospital, they will either receive one dose of saline solution via their NG tube plus non-surgical management (Control arm) or one dose of Gastrografin via their NG tube plus non-surgical management (Gastrografin arm). At any point during the study if the patient's clinical condition changes and the surgical team thinks the patient needs an operation then it will occur regardless of enrollment in the study.

Prior to the patient receiving Gastrografin or saline solution, the investigators will confirm that the patient does not have an allergy to iodine, as Gastrografin contains high levels of iodine, and that they have normal thyroid hormone levels. The investigators will test the patient's levels of thyroxine (T4) and thyroid stimulating hormone (TSH) by blood draw, as excessive iodine exposure can block thyroid hormone synthesis in young children. The investigators will be able to test thyroid hormone levels from the patients initial blood work at admission, which occurs as part of the patient's standard care. This way there will be no delay in the treatment of the small bowel obstruction (SBO) due to waiting for lab results and the patient can receive either treatment at 24 hours post admission. Thyroid hormone levels will be tested throughout the study for the Gastrografin group from routine blood draws that are part of standard care when a patient is NPO. Therefore no additional blood draws will be required as part of the study. If the patient's thyroid hormone levels are normal they can be enrolled in the study. If not, they will not be eligible to participate in the study.

Twenty-four hours following admission and consent, patients will either receive Gastrografin or an equivalent volume of saline (Control arm) via the NG tube, depending on the arm offered at their centre. In both cases, the NG tube will be clamped for 30 minutes to one hour. Doses of Gastrografin will be proportional to the patient's age and will be based on the recommendations from the manufacturer (i.e., product monograph) and published studies. Dosages will range from 30ml for children up to 5 year of age to 60ml for children between 5-18 years and will not be diluted. The manufacturer only recommends diluting Gastrografin if the patient is of low-birth weight or is considered debilitated. Since none of the patient recruited for this study will meet these criteria, Gastrografin will not be diluted. Patients who do not receive Gastrografin will receive an equivalent volume of saline solution via the NG tube in addition to non-surgical management, which includes NG tube decompression, NPO, and IV fluids. At this time (24 hours post admission) an x-ray will be completed for both study arms.

After the patient receives Gastrografin or saline solution they will continue to be monitored for the duration of the study. The patients in both groups will receive an abdominal x-ray at 12 hours after they have been given Gastrografin or saline (36 hours since admission). If Gastrografin is present in the cecum, feeding will be initiated and the patient will be observed closely to monitor the success of Gastrografin administration. If not viewed at 12 hours post administration, non-surgical management will be maintained until resolution of the bowel obstruction or surgical intervention. Standard procedure for initiating feeds will be used on all children included in the study. The initiation of feeding is up to the discretion of the attending paediatric surgeon and is typically determined based on resolution of the bowel obstruction, decrease in NG tube drainage, the degree of abdominal distension, and the passage of stool. Patients given saline via the NG tube as part of the Control arm will also receive an x-ray at 12 hours post saline solution and will continue to receive non-surgical management until resolution or surgical intervention.

The data collection period is from admission to discharge; there will be no data collection at any follow-up appointment. Patients will be seen in clinic for follow-up post SBO at the discretion of the attending surgeon and this will not differ based on study group (Gastrografin vs. Control). The majority of the information will be collected from the patient's chart and will not require directly consulting with the patient or their parents/caregivers. In order to have an equal number of patients in each group, the investigators will set a cap of 73 patients per group. Once one of the study arms reaches 73 patients, the investigators will stop enrolling into that arm of the study and only offer the other arm to potential patients. This will help to ensure that the expected sample is achieved in each group and that groups are not uneven. Enrollment rate are expected to be fairly even between study arms, as the treatment arm is non-invasive, has a strong body of evidence around its effectiveness in other conditions, and has a very low complication rate. Additionally, the fact that it is being used outside of the study at the participating centres at the discretion of the paediatric surgeons may provide an added level of reassurance for the patient and their family.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed small bowel obstruction by a surgeon or physician
* Patient has undergo 24 hours of monitoring and non-surgical management (NG tube decompression, IV fluids, and NPO)
* Patients are between 6 month and 18 years of age at time of diagnosis

Exclusion Criteria:

* Abnormal levels of thyroid stimulating hormone (TSH) or thyroxine (T4)
* Prior thyroid surgery
* Receiving thyroid hormone replacement therapy
* Allergy to medical or non-medial ingredients in Gastrografin
* Weight of less than 10kg at time of diagnosis

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
rate of surgical intervention | Through study completion, up to 6 months
  number of patients who require surgical intervention to resolve their bowel obstruction after receiving either treatment.

SECONDARY OUTCOMES:
Length of hospital stay | Through study completion, up to 6 months
  The length of time the patient was admitted to the hospital for the treatment of their small bowel obstruction
Time to first feed | Through study completion, up to 6 months
  Since patients are NPO at admission, this will capture the length of time from admission to when the patient is first given oral feeds
Time to full feeds | Through study completion, up to 6 months
  Since patients are NPO at admission, this will capture the length of time from admission to when the patient consistently reaches their targeted caloric intake.
Rate of complications | Through study completion, up to 6 months
  Capture all Gastrografin-specific and other complications related to their hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital, London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Background] Moss RL, Henry MC, Dimmitt RA, Rangel S, Geraghty N, Skarsgard ED. The role of prospective randomized clinical trials in pediatric surgery: state of the art? J Pediatr Surg. 2001 Aug;36(8):1182-6. doi: 10.1053/jpsu.2001.25749. PMID 11479852
- [Background] Rangel SJ, Narasimhan B, Geraghty N, Moss RL. Development of an internet-based protocol to facilitate randomized clinical trials in pediatric surgery. J Pediatr Surg. 2002 Jul;37(7):990-4; discussion 990-4. doi: 10.1053/jpsu.2002.33826. PMID 12077756
- [Background] St-Louis E, Oosenbrug M, Landry T, Baird R. Enrollment and reporting practices in pediatric general surgical randomized clinical trials: A systematic review and observational analysis. J Pediatr Surg. 2018 May;53(5):879-884. doi: 10.1016/j.jpedsurg.2018.02.009. Epub 2018 Feb 8. PMID 29501236
- [Background] Ahmet A, Lawson ML, Babyn P, Tricco AC. Hypothyroidism in neonates post-iodinated contrast media: a systematic review. Acta Paediatr. 2009 Oct;98(10):1568-74. doi: 10.1111/j.1651-2227.2009.01412.x. Epub 2009 Jul 3. PMID 19575766
- [Derived] Emil S, Guadagno E, Baird R, Puligandla P, Romao R, Van HouWelingen L, Yanchar NL; Canadian Consortium for Research in Pediatric Surgery (CanCORPS). The Canadian Consortium for Research in Pediatric Surgery: Roadmap for Creation and Implementation of a National Subspecialty Research Consortium. J Am Coll Surg. 2022 Dec 1;235(6):952-961. doi: 10.1097/XCS.0000000000000396. Epub 2022 Nov 15. PMID 36102499